CLINICAL TRIAL: NCT03027869
Title: Normal Brain Imaging Database for Brain Disorder Studies
Acronym: Normal_tDCS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Ji Hyun Ko, PhD, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B2016:074
Record Dates: First submitted 2017-01-16; First posted 2017-01-23 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Real Left DLPFC tDCS (Active Comparator): Real tDCS on the left dorsolateral prefrontal cortex
  Interventions: Device: transcranial direct current stimulation
- Sham tDCS (Sham Comparator): 30sec ramp-up and 30sec ramp-down
  Interventions: Device: transcranial direct current stimulation
- Real Right DLPFC tDCS (Active Comparator): Real tDCS on the right dorsolateral prefrontal cortex
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — 15 minute anodal stimulation 1.5mA

SUMMARY:
Healthy volunteers will be recruited. All subjects will be tested a battery of neuropsychological tests, then undergo fluorodeoxyglucose-positron emission tomography (PET) and magnetic resonance imaging (MRI). During the PET and MRI, they will be stimulated with transcranial direct current stimulation (tDCS) for 15 minutes. A third of subjects will receive real tDCS on the left prefrontal cortex, a third on the right prefrontal cortex, and the other third will receive sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* N/A

Exclusion Criteria:

* History of any neurological or psychiatric diseases;
* Abnormal MRI;
* metal implants or a cardiac pacemaker;
* Pregnant or breastfeeding women (female subjects of child bearing potential will be screened for pregnancy before MRI imaging).
* severe hypertension.
* cardiovascular disease.
* Family history of epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-28 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
functional connectivity | immediate (less than 30 minutes)
  The functional connectivity of the right caudate nucleus will be estimated using graph theory analysis technique of resting-state fMRI.

SECONDARY OUTCOMES:
Stroop task performance | immediate (less than 60 minutes)
  the executive function that is thought to involve the caudate nucleus will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No